CLINICAL TRIAL: NCT05081362
Title: Cardiovascular Assessment in Patient Recovered From COVID-19 and Recovery of Autonomic Nervous System in Association With the Severity of the Disease
Acronym: COVIDans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Head of cardiovascular anesthesiology and intensive care, IRCCS Policlinico S. Donato
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COVIDans
Record Dates: First submitted 2021-10-07; First posted 2021-10-18 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — epicatechin gallate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COVID-severe (Other): patient recovered from severe COVID desease
  Interventions: Other: Non invasive cardiovascular monitoring with CNAP device of arterial pressure, ECG and respiratory activity
- COVID-moderate (Other): patient recovered from moderate COVID desease
  Interventions: Other: Non invasive cardiovascular monitoring with CNAP device of arterial pressure, ECG and respiratory activity
- COVID-mild (Other): patient recovered from mild COVID desease
  Interventions: Other: Non invasive cardiovascular monitoring with CNAP device of arterial pressure, ECG and respiratory activity

INTERVENTIONS:
Other: Non invasive cardiovascular monitoring with CNAP device of arterial pressure, ECG and respiratory activity — Non invasive cardiovascular monitoring with CNAP device of arterial pressure, ECG and respiratory activity during ten minutes in rest and ten minutes in orthostatic position

SUMMARY:
The goal of the study is to assess autonomic nervous system and cardiovascular controll during orthostatic challenge in 90 patients recovered from COVID-19 and devided into three groups depend on severity of the morbidity.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* spontaneous sinus rhythm
* signed informed consent

Exclusion Criteria:

* no spontaneous sinus rhythm
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Arterial pressure measured in mmHg | 6 months
  Continuous measurement of the arterial pressure for 10 minutes in rest and 10 minutes in orthostatic position.
Heart rate measured in bpm | 6 months
  Continuous measurement of heart rate for 10 minutes in rest and 10 minutes in orthostatic position.
Respiratory frequency | 6 months
  Continuous measurement of respiratory frequency for 10 minutes in rest and 10 minutes in orthostatic position.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No